CLINICAL TRIAL: NCT02144441
Title: Proof-of-concept Trial of Clinician-supported Patient Self-management of Hospital Insulin Therapy
Brief Title: Pilot Study of Clinician-supported Patient Self-management of Hospital Insulin Therapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Very few patients met eligibility criteria, none of whom elected to enroll.
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 819840
Record Dates: First submitted 2014-05-13; First posted 2014-05-22 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2014-05

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; Insulin; Self Administration; Patient Satisfaction; Glucose; Hypoglycemia; Hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance; Patient Satisfaction; Hypoglycemia; Hyperglycemia | interventions — Insulin Glargine; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patient self-administered insulin (Experimental): The study's only arm
  Interventions: Drug: glargine and aspart

INTERVENTIONS:
Drug: glargine and aspart — Inpatient will administer hospital-dispensed basal-bolus insulin (glargine and aspart) according to a regimen developed in collaboration with the diabetes consult service.

SUMMARY:
This study will examine the feasibility of implementing a clinician-supported patient self-managed inpatient insulin intervention. It will: assess the number of eligible patients presenting over time; assess patients' willingness to enroll; assess patients' ability to successfully complete the intervention; examine occurrences of hyperglycemia and hypoglycemia; and assess patients' satisfaction with inpatient diabetes care.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the Hospital of the University of Pennsylvania (HUP) in the past 72 hours.
* Current HUP locations are Founders 12, Founders 14, Silverstein 11, and Rhoads 1.
* Age 18 years or older.
* Type-1 or type-2 diabetes mellitus requiring home basal-bolus insulin therapy administered via subcutaneous injection (not pump).
* Patient manages own basal-bolus insulin therapy at home without assistance, including measuring own blood glucose (at least at mealtimes) and administering own subcutaneous insulin.
* Patient is willing to use the following insulin products: rapid-acting insulin aspart via insulin pen (NovoLog) and long-acting insulin glargine via vial and syringe (Lantus).
* Most recent hemoglobin A1c was measured within past 6 months and was <7.5%.
* Active order for in-hospital basal-bolus or sliding-scale insulin.
* Patient is willing and able to record their self-measured blood glucose results, doses of insulin that they self-administer, a food journal, and exercise log.
* Clinical care team agrees with study inclusion.

Exclusion Criteria:

* Inpatient order for insulin via subcutaneous infusion (i.e., pump) or intravenous infusion (i.e., drip).
* Inability to perform the activities required by the trial.
* Primary reason for admission was hyperglycemia, hypoglycemia, diabetic ketoacidosis, hyperglycemic hyperosmolar nonketotic coma, a psychiatric condition, acute alcohol poisoning, or acute drug ingestion.
* Order for a newly-prescribed or increased dose of a previously-prescribed corticosteroid.
* Enteral or parenteral nutrition.
* Expected length of stay <48h, as determined by treating physician.
* At risk for self-harm, as determined by 1-to-1 status placement.
* Pregnant, as recorded on medical record.
* Cannot understand, speak, and read English.
* Patient does not wish to utilize Novolog and Lantus while in the hospital.
* Prior enrollment in this trial.
* Do not resuscitate status.
* Inability to give written informed consent.
* Clinical care team disagrees with study inclusion.
* Patient has limited mobility such that they cannot safely access the bedside medication lockbox.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Trial feasibility metric: number of screened patients | 3 months
Trial feasibility metric: number of eligible patients | 3 months
Trial feasibility metric: number of patients approached for consent | 3 months
Trial feasibility metric: proportion of eligible patients not consenting | 3 months
Trial feasibility metric: reasons for non-consent | 3 months
Trial feasibility metric: characteristics of consenting subjects and non-consenting patients | 3 months
  To examine baseline demographics and clinical factors, such as: mean age, median age, proportion female sex, other demographics, proportion with type I diabetes, proportion with type II diabetes, hemoglobin A1c on admission, reasons for admission
Trial feasibility metric: proportion of enrolled subjects completing the intervention | 3 months
Trial feasibility metric: proportion of enrolled subjects disenrolling | 3 months
Trial feasibility metric: reasons for disenrollment | 3 months

SECONDARY OUTCOMES:
Hyperglycemia | During hospitalization (maximum length 7 days)
  Frequency of blood glucose concentrations that are hyperglycemic (> 180 mg/dL)
Patient satisfaction | At the end of hospitalization (maximum length 7 days)
  Satisfaction with inpatient diabetes care, as measured by the Diabetes Treatment Satisfaction Questionnaire for Inpatients (DTSQ-IP) adapted for use in the United States
Hypoglycemia | During hospitalization (maximum length 7 days)
  Frequency of hypoglycemia (blood glucose concentration < 70 mg/dL) and frequency of severe hypoglycemia (blood glucose concentration < 40 mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Sean Hennessy, PharmD, PhD, Principal Investigator — Perelman School of Medicine at the University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Acton EK, Leonard CE, Schutta MH, Cardillo S, Troxel AB, Trotta R, Hennessy S. Challenges in recruiting subjects to a pilot trial of patient-managed in-hospital insulin. BMC Res Notes. 2015 Oct 1;8:523. doi: 10.1186/s13104-015-1480-6. PMID 26429339